CLINICAL TRIAL: NCT05050149
Title: A Multicenter, Phase 2, Open-Label Study Evaluating The Safety And Efficacy of Sirolimus 3.9% Topical Gel (PTX-022) In The Treatment of Microcystic Lymphatic Malformations
Brief Title: Study Evaluating the Safety and Efficacy of PTX-022 (QTORIN Sirolimus) in the Treatment of Microcystic Lymphatic Malformations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Palvella Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PALV-06
Record Dates: First submitted 2021-09-08; First posted 2021-09-20 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Microcystic Lymphatic Malformation
MeSH Terms: conditions — Lymphangioma

STUDY DESIGN:
Intervention Model Description: This is an open-label, baseline-controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: PTX-022 (Experimental): PTX-022 QTORIN
  Interventions: Drug: PTX-022

INTERVENTIONS:
Drug: PTX-022 — Safety and Efficacy of PTX-022 in the Treatment of Microcystic Lymphatic Malformations

SUMMARY:
This study evaluates the safety and efficacy of PTX-022 (sirolimus) Topical Gel 3.9% w/w in the treatment of Microcystic Lymphatic Malformations. The participant will receive 3 months of PTX-022 treatment by the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 6 years or older
* Diagnosed with Microcystic Lymphatic Malformations
* Able and willing to comply with all protocol-required activities
* Willing and able to provide written informed consent

Exclusion Criteria:

* Any significant concurrent condition that could adversely affect participation.
* Any history of allergy or hypersensitivity to sirolimus, or sirolimus-like medications or to PTX-022
* Patient's deemed by the investigator as unwilling or unable to remain compliant with all tests and procedures, including adherence to study drug administration and other protocol-required activities.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Stanford University, Palo Alto, California
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Vascular Birthmark Institute, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Pennsylvania (CHOP), Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teng JMC, Hammill A, Martini J, Treat J. Sirolimus in the Treatment of Microcystic Lymphatic Malformations: A Systematic Review. Lymphat Res Biol. 2023 Apr;21(2):101-110. doi: 10.1089/lrb.2021.0103. Epub 2022 Jul 18. PMID 35852876

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental: PTX-022
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: PTX-022
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (13.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0
  Race: Asian | 1
  Race: Black or African American | 2
  Race: Native Hawaiian or Other Pacific Islander | 0
  Race: White | 8
  Race: Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events
Time Frame: 4 months
Measure: Number; unit: participants
Arm/Group | Experimental: PTX-022
Number analyzed (Participants) | 12
participants
  Subjects with TEAEs | 9
  Gastrointestinal Disorders | 2
  General Disorders and Administration Site Conditions | 6
  Infections and Infestations | 2
  Investigations | 1
  Musculoskeletal and Connective tissue Disorders | 1
  Nervous System Disorders | 2
  Renal and Urinary Disorders | 1
  Skin and Subcutaneous Tissue Disorders | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from screening until Month 4
Arm/Group | Experimental: PTX-022
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 9/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: PTX-022 (N=12)
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Application Site Discharge (General disorders) | 1
Application Site Erythema (General disorders) | 1
Application Site Pain (General disorders) | 3
Application Site Paraesthesia (General disorders) | 1
Application Site Pruritus (General disorders) | 3
Nodule (General disorders) | 1
Folliculitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Reticulocyte count increased (Investigations) | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Micturition urgency (Renal and urinary disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/49/NCT05050149/Prot_SAP_000.pdf